CLINICAL TRIAL: NCT06264921
Title: A Phase 1, First-in-Human, Open-Label Study to Evaluate the Safety, Tolerability, PK, and Preliminary Anti-tumor Activity of the Novel Orally Available CDK2 Inhibitor NKT3447 in Adults With Advanced/Metastatic Solid Tumors
Brief Title: A Study With NKT3447 for Adults With Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated as a result of Sponsor portfolio reprioritization.
Sponsor: NiKang Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NKT3447-101
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Solid Tumor, Adult; Advanced Solid Tumor; Metastatic Tumor; Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Metastatic Ovarian Carcinoma; Endometrial Cancer; Endometrial Neoplasms; Endometrial Diseases; Metastatic Endometrial Cancer; Metastatic Endometrial Carcinoma; Advanced Endometrial Carcinoma; Advanced Ovarian Carcinoma; Gastric Cancer; Advanced Gastric Carcinoma; Metastatic Gastric Cancer; Metastatic Gastric Carcinoma; Small-cell Lung Cancer; Small Cell Lung Carcinoma; Triple Negative Breast Cancer; Triple Negative Breast Neoplasms; Platinum-resistant Ovarian Cancer; Platinum-refractory Ovarian Carcinoma; CCNE1 Amplification; Hormone Receptor Negative Breast Carcinoma; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Progesterone-receptor-positive Breast Cancer
Keywords: CDK 2 Inhibitor; CDK 4 Inhibitor; CDK 6 Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Diseases; Stomach Neoplasms; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Dose Expansion
Masking Description: Randomized for the Expansion Phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation will assess the safety, efficacy, and PK/PD data of oral dosing NKT3447 at increasing dosage levels to determine the MTD and/or preliminary RDEs.
  Interventions: Drug: NKT3447
- Dose Expansion (Experimental): Dose expansion will include 2 RDEs selected to determine the preliminary antitumor activity and the RP2D.
  Interventions: Drug: NKT3447

INTERVENTIONS:
Drug: NKT3447 — Oral CDK2 inhibitor

SUMMARY:
The goal of the Dose Escalation phase of the study is to evaluate the safety, tolerability, and pharmacokinetics (PK) to determine the maximum tolerated dose (MTD) and/or preliminary recommended dose for expansion (RDE) of NKT3447 in adults with advanced or metastatic solid tumors. The goal of the Expansion phase of the study is to evaluate the safety, tolerability, pharmacokinetics (PK), and the preliminary antitumor activity of NKT3447 in adult subjects with cyclin E1 (CCNE1) amplified ovarian cancer at the RDEs selected in Dose Escalation and to determine the preliminary recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This is a Phase 1/1b, first-in-human, open-label, multicenter study of NKT3447 in adults with advanced/ metastatic solid tumors. The study consists of 2 parts, a Dose Escalation phase and a Dose Expansion phase. Eligible patients must have confirmed advanced/metastatic solid tumors (as outlined below) with disease progression on prior standard treatment, intolerance to or ineligibility for standard treatment, or no available standard treatment likely to improve the disease outcome in the judgment of the investigator.

Dose Escalation:

1. Ovarian cancer
2. Endometrial cancer
3. Gastric cancer or gastroesophageal junction cancer
4. Small cell lung cancer
5. Triple-negative breast cancer (human epidermal growth factor receptor 2, estrogen receptor, progesterone receptor negative)
6. Estrogen receptor/progesterone-receptor positive (ER+/PR+), human epidermal growth factor receptor 2 negative (HER2-) breast cancer (must have progressed following treatment with a CDK4/6 inhibitor, and not suitable for endocrine therapy)
7. Other solid tumors with CCNE1 amplification as determined by next generation sequencing by local liquid or tissue biopsy.

Dose Expansion:

a. Platinum resistant or refractory ovarian cancer (defined as recurrence ≤6 months after completing platinum-based regimen) with progression on at least 1 platinum containing therapy with cyclin E amplification as determined by fluorescence in situ hybridization, quantitative polymerase chain reaction, or next-generation sequencing by local liquid or tissue biopsy.

The Dose Escalation phase will evaluate the safety, tolerability, and pharmacokinetics (PK) to determine the maximum tolerated dose (MTD) and/or preliminary recommended dose for expansion (RDE) of NKT3447 in adults with advanced or metastatic solid tumors.

The Dose Expansion phase will evaluate the safety, tolerability, pharmacokinetics (PK), and the preliminary antitumor activity of NKT3447 in adult subjects with CCNE1 amplified ovarian cancer at the RDEs selected in Dose Escalation and to determine the preliminary recommended RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed unresectable advanced/metastatic solid tumors (as outlined below) with disease progression on prior standard treatment, intolerance to or ineligibility for standard treatment, or no available standard treatment likely to improve the disease outcome in the judgment of the Investigator.

  * Measurable disease per the RECIST v1.1
  * An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
  * Able to swallow oral medications.

Dose Escalation(Part 1):

1. Ovarian cancer
2. Endometrial cancer
3. Gastric cancer or gastroesophageal junction cancer
4. Small cell lung cancer (SCLC)
5. Triple-negative breast cancer (human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], progesterone receptor negative)
6. ER/progesterone-receptor positive, HER2 negative breast cancer (must have progressed following treatment with a CDK4/6 inhibitor, and not suitable for endocrine therapy)
7. Other solid tumors with CCNE1 amplification as determined by NGS by local liquid or tissue biopsy.

Dose Expansion (Part 2):

a. Platinum resistant or refractory ovarian cancer (defined as recurrence ≤6 months after completing platinum-based regimen) with progression on at least 1 platinum containing therapy with CCNE1 amplification as determined by NGS by local liquid or tissue biopsy.

* Measurable disease per the RECIST v1.1
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Able to swallow oral medications.

Exclusion Criteria:

* Locally advanced solid tumor that is a candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
* History of another malignancy with exceptions
* Visceral crisis with life-threatening complications, lymphangitic spread, CNS metastasis and/or carcinomatous meningitis
* Failed to recover from effects of prior anticancer treatment therapy to baseline or Grade ≤ 1 severity (per CTCAE)
* Clinically active interstitial lung disease
* History of uveitis, retinopathy or other clinically significant retinal disease
* Has known human immunodeficiency virus (HIV), active hepatitis B or C infection
* Prior CDK2 inhibitor
* Major surgery within 2 months or minor surgery within 10 days before the first dose of NKT3447

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) events | 28 days
  DLTs graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5 .0.
Objective Response Rate (ORR) | 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as determined by the Investigator

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of disease progression or death.
Duration of Response (DOR) | 2 years
  Duration of overall response is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.
Disease control rate | 1 year
  Disease control rate defined as CR + PR + stable disease [SD]
Overall Survival (OS) | 2 years
  OS defined as the time from the date the participant started study drug to death for any reason.
Time to Response (TTR) | 1 year
  TTR is defined as the time from first dose to the first documented CR or PR which is subsequently confirmed.
Number of Participants with Adverse Events | 2 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
Maximum observed plasma concentration (Cmax) of NKT3447 | 1 month
  Maximum observed plasma concentration (Cmax) of NKT3447
Time to maximum observed plasma concentration of NKT3447 (Tmax) | 1 month
  Time to maximum observed plasma concentration of NKT3447 (Tmax)
Observed trough concentration of NKT3447 (Ctrough) | 88 weeks
  Observed trough concentration of NKT3447 (Ctrough)
Area under the plasma concentration-time curve (AUC0-t) of NKT3447 | 1 month
  Area under the plasma concentration-time curve (AUC0-t) of NKT3447
Apparent clearance (CL/F) | 1 month
  Apparent clearance (CL/F)
Apparent volume of distribution (V/F) | 1 month
  Apparent volume of distribution (V/F)
Half-life (t1/2) | 1 month
  Half-life (t1/2)
Accumulation ratio (AR) | 1 month
  Accumulation ratio (AR)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - AdventHealth Cancer Institute, Celebration, Florida
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Norton Cancer Institute - Broadway, Louisville, Kentucky
  - The Gabrail Pharmacology Phase 1 Research Center, Canton, Ohio
  - Texas Oncology-Austin Midtown NEXT Oncology, Austin, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared at this time